CLINICAL TRIAL: NCT02682212
Title: Obstetric Perineal Trauma, Pelvic Floor Symptoms and Early Physiotherapy Intervention
Brief Title: Obstetric Perineal Trauma and Physiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landspitali University Hospital (Other)
Collaborators: University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LSH-15-001
Record Dates: First submitted 2015-03-30; First posted 2016-02-15 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy Complications
Keywords: Pelvic floor; obstetrics; perineal tear; physiotherapy
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy intervention (Experimental): Intensive pelvic floor muscle training (PFMT) given by a physiotherapist with vaginal/rectal pressure feedback once a week for 12 weeks.
  Interventions: Other: Physiotherapy intervention
- No intervention (No Intervention): Standard care

INTERVENTIONS:
Other: Physiotherapy intervention — Compare the effect of early physiotherapy intervention (pelvic floor muscle training, PFMT) with standard care on pelvic floor dysfunction symptoms, quality of life (QoL) and (pelvic floor muscle (PFM) strength, for women who answered the questionnaire positively for 1) urinary incontinence, 2) other dysfunction of the pelvic floor.
  Arms: Physiotherapy intervention

SUMMARY:
The main objective is to investigate effects of perineal trauma at birth on women´s health and whether early physiotherapy improves pelvic floor strength. This will be achieved by an acknowledged/validated questionnaire sent electronically 6 weeks after first delivery. Women with symptomes of urinary incontinence according to the questionnaire will be offered participation in a single-blinded randomized intervention study to compare outcome after targeted physiotherapy with conventional advice and support. Intervention encompasses weekly pelvic floor training for 12 weeks. Pelvic strength will be measured and symptom information collected before and after intervention and 12 months postpartum in both groups.

Pelvic floor problems after delivery are common and often persistent, including urinary/fecal incontinence, pelvic organ prolapse and sexual problems. Such symptoms reduce QoL and handicap women in multiple ways, physically, psychologically and socially. More knowledge of whether interventions and guidelines in this field can improve health and QoL is required.

DETAILED DESCRIPTION:
Single-blind randomized controlled trial (RCT) to assess and compare the effects of early pelvic floor muscle training and present standard care/advice on pelvic floor muscle (PFM) strength, symptoms from the pelvic floor and bothersome symptoms (QoL) after obstetric perineal repair.

Procedure/Study design: Single-blind randomized controlled trial.

Details of test administration and data collection methods:

PFM strength will be measured with Myomed 932® (Enraf-Nonius, Delft, Netherlands) for squeeze pressure, vaginally and rectally.

Pelvic floor symptoms, (bladder/bowel function, prolapse symptoms, sexual function) and bothersomeness will be measured with the validated Icelandic version of the Australian Female Pelvic Floor Questionnaire.

Assessment and treatment will begin from 6th week postpartum. After initial assessment, instruction on pelvic floor function the pelvic floor questionnaire administration, participants will be randomized to intervention and control groups by a person not involved in measurements or treatment. The intervention group will receive individual treatment by a physiotherapist not involved in the initial assesment. This will be in the form of intensive PFMT with vaginal/rectal pressure feedback once a week for 12 weeks and be encouraged to do daily exercises. Repeated assessment of pelvic floor function and questionnaire administration will be after 12 weeks for both groups and repeated 12 months after birth.

Assessment of pelvic floor function includes rectal/vaginal resting pressure, PFM strength (maximal voluntary contraction, strongest of three measured as a vaginal and anal squeeze pressure), and endurance for 10 sec (area under the curve both rectal and vaginal).

Preliminary assumption of power (beta) of 80% and a level of significance (alfa) of 5% and estimating 1 against 3 women with symptoms of urinary incontinence in treatment vs. control groups, respectively after intervention, ca. 40 women will be needed per group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy primiparas after delivery at LSH
* ≥18 years
* Diagnosed with urinary incontinence according to the self administered Australian Pelvic floor Questionnaire (Icelandic version) 6 weeks post partum.
* Able to attend intervention in the capital area
* Answer the Australian Pelvic Floor Questionnaire

Exclusion Criteria:

* Diseases or conditions that can interfere with pelvic floor function (other than childbirth), such as prior pelvic floor surgery or ability to benefit from the intervention
* Women unable to understand Icelandic
* Woman with cognitive disabilities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence rates measured by scores on the Australian Female PelvicFloor questionnaire | 16 weeks
  Urinary incontinence rates measured by scores on the Australian Female PelvicFloor questionnaire

SECONDARY OUTCOMES:
Fecal/flatal incontinence measured by scores on the Australian Female PelvicFloor questionnaire | 16 weeks
  Fecal/flatal incontinence measured by scores on the Australian Female PelvicFloor questionnaire
Sexual dysfunction measured by scores on the Australian Female PelvicFloor questionnaire | 16 weeks
  Sexual dysfunction measured by scores on the Australian Female PelvicFloor questionnaire
Quality of life measured by scores on the Australian Female PelvicFloor questionnaire | 16 weeks
  Quality of life measured by scores on the Australian Female PelvicFloor questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thora Steingrimsdottir, MD, PhD, Principal Investigator — Landspitali University Hospital/University of Iceland, Reykjavik, Iceland; Kari Bo, PhD, Study Chair — Norwegian School of Sports Sciences, Oslo, Norway
Locations (1):
- Tap, Physical Therapy Clinic, Kopavogur, Iceland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Sigurdardottir T, Steingrimsdottir T, Geirsson RT, Halldorsson TI, Aspelund T, Bo K. Can postpartum pelvic floor muscle training reduce urinary and anal incontinence?: An assessor-blinded randomized controlled trial. Am J Obstet Gynecol. 2020 Mar;222(3):247.e1-247.e8. doi: 10.1016/j.ajog.2019.09.011. Epub 2019 Sep 14. PMID 31526791